CLINICAL TRIAL: NCT02763917
Title: AIRWEIGHS: Investigating Obesity as a Susceptibility Factor for Air Pollution in Childhood Asthma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: IRB00074171; P50ES018176 (NIH)
Record Dates: First submitted 2016-05-03; First posted 2016-05-05 (Estimated); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Air Purifier (Active Comparator): Two portable air purifiers containing HEPA filters will be placed in the bedroom and room where the participant reports spending the most time. We have chosen to deploy two air purifiers because we have observed a 50% reduction in indoor PM concentrations with two air purifiers. Participants will be instructed to run the air purifiers continually. Participants will receive educational materials about environmental factors that are important for asthma health and environmental modification strategies. Participants will also receive educational materials about health benefits of maintaining a normal weight.
  Interventions: Device: Active Air Purifier
- Placebo Air Purifier (Placebo Comparator): Homes in the control group will receive placebo air purifiers that have the internal air filters removed, but which will run normally. Participants will receive educational materials about environmental factors that are important for asthma health and environmental modification strategies, and educational materials about health benefits of maintaining a normal weight. At the end of the study, participants in the control group will receive active air purifiers. A control group is needed to ensure that reduced pollutant levels and health effects are not due to temporal trends and 'placebo effects' of being enrolled in an intervention trial. Participants will also be informed that being in the study does not prevent them from purchasing and using air cleaners during the study period.
  Interventions: Device: Placebo Air Purifier

INTERVENTIONS:
Device: Active Air Purifier — Two portable air purifiers containing HEPA filters will be placed in the bedroom and room where the participant reports spending the most time. Participants will be instructed to run the air purifiers continually. Participants will receive educational materials about environmental factors that are important for asthma health and environmental modification strategies, and educational materials about health benefits of maintaining a normal weight.
  Arms: Active Air Purifier
Device: Placebo Air Purifier — Homes in the control group will receive placebo air purifiers that have the internal air filters removed, but which will run normally. Participants will receive educational materials about environmental factors that are important for asthma health and environmental modification strategies, and educational materials about health benefits of maintaining a normal weight. At the end of the study, participants in the control group will receive active air purifiers. A control group is needed to ensure that reduced pollutant levels and health effects are not due to temporal trends and 'placebo effects' of being enrolled in an intervention trial. Participants will be informed that being in the study does not prevent them from purchasing and using air cleaners during the study period.
  Arms: Placebo Air Purifier

SUMMARY:
Background: Asthma and obesity are public health crises that have concurrently risen over the past decades, affecting millions of children in the United States and disproportionately affecting low-income minority children in urban areas. The same children at highest risk for asthma and obesity also have greater exposure to indoor and outdoor pollution. Emerging evidence suggests that obesity may confer increased susceptibility to health effects of air pollution.

Methods: Aiming to provide causal-level evidence of these observational findings, we propose a home intervention study to 1) test whether targeted reductions of indoor Particulate Matter (PM) concentrations improve the respiratory health of overweight inner-city children with asthma more than that of lean inner-city children with asthma and 2) investigate mediators of susceptibility to indoor PM among overweight versus lean children with asthma. We will accomplish these aims using a 1:1 randomized controlled trial of 200 children with persistent asthma (half normal weight, half overweight) living in Baltimore City. Participants will be randomized to receive either two active air purifiers containing high-efficiency particulate air (HEPA) filters or two sham air purifiers with their filters removed.

Implications: If the aforementioned observational findings are confirmed, implications will be directly relevant to the over 170 million children around the world now estimated to be overweight or obese.

DETAILED DESCRIPTION:
The primary object of this study is to determine the efficacy of a targeted environmental intervention among overweight inner city children as compared to normal weight inner city children with asthma.

Specific Aim #1: To determine if overweight inner-city children, compared to lean inner-city children, have greater improvement in asthma with an air purifier intervention aimed at reducing indoor PM.

Hypothesis 1: An intervention using HEPA filter air purifiers in the homes of inner-city children with asthma will be associated with greater respiratory improvement in overweight children than in normal weight children.

Specific Aim #2a: To investigate mediators of susceptibility among overweight versus normal weight children with asthma.

Hypothesis #2. Candidate mediators, including increases in a) tidal volume and thereby increases in doses of inhaled particles, b) inflammatory and oxidative stress responses, c) corticosteroid resistance, and d) sleep disordered breathing mediate increased susceptibility to indoor PM among overweight versus normal weight children with asthma.

Children with asthma will be enrolled in the study for about 16 weeks. They will have three clinic visits, an overnight sleep study, and two home environmental assessments for one week each. They will have a home and clinical assessment before randomization and another home and clinical assessment about 12 weeks after randomization. The primary outcome measure is maximum number of asthma symptom days.

ELIGIBILITY:
Inclusion Criteria:

1. 8-17 years of age
2. Persistent asthma (NAEPP criteria)
3. Exacerbation in previous 12 months
4. Non-smoker
5. Spends ≥4 nights/week at home
6. No plans to move during the study

Exclusion Criteria:

1. Significant pulmonary or cardiac disease
2. Home not appropriate candidate due to disrepair
3. Underweight, defined by BMI <5th percentile
4. Pregnancy

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 198 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Maximum Symptom Days | Baseline and about 12 weeks after the intervention
  We have chosen symptoms based on the strong relationship between symptoms and PM observed in previous studies. Symptoms during the previous two weeks will be captured with standardized questions used in many inner-city asthma studies, including our own that detected a strong association between indoor PM and asthma symptoms. A 'maximum symptom days' variable will constructed as the maximum of the variables: days of slowed activity, days of wheezing, coughing or chest tightness when running or going upstairs, and nights of waking with asthma symptoms in the past two weeks. We will administer questionnaires to the primary caregiver of children 8-11 years and to both participant and caregiver for adolescents age 12-17. Previous studies have indicated concordance between adolescent and the caregiver responses, and we will collect data to assess concordance within our study population. Individual symptom variables will serve as secondary outcomes.

SECONDARY OUTCOMES:
Asthma Control | Baseline and about 12 weeks after the intervention
  Asthma Control Questionnaire (ACT). This questionnaire assesses asthma control and a score of less than 19 has been linked to poor asthma control. The Asthma Therapy Assessment Questionnaire includes questions about asthma control and will also be used.
Asthma Symptoms | Baseline and about 12 weeks after the intervention
  The Asthma Symptom Utility Index (ASUI) will be used to assess asthma symptoms.
Health Care Utilization | Baseline and about 12 weeks after the intervention
  Child participants and caregivers will be asked about acute health care encounters during the study, including unscheduled doctor visits, Emergency Department visits, and hospitalizations. Acute visits occurred in approximately 30% of our previous study populations during a 3 month period.
Lung Function | Baseline and about 12 weeks after the intervention.
  Pre- and post-bronchodilator forced expiratory vital capacity in the first second/forced vital capacity (FEV1/FVC) and FEV1 will be measured and interpreted according to the American Thoracis Society (ATS) guidelines using NHANES predicted equations.
FENO | Baseline and about 12 weeks after the intervention
  Exhaled nitric oxide (FENO) will provide a non-invasive means of assessing pulmonary inflammation in a large cohort of children. Measurements will be obtained prior to lung function according to the American Thoracic Society Guidelines with handheld, FDA-approved analyzer (NIOX System, Aerocrine, Sweden)

CONTACTS AND LOCATIONS:
Overall Officials: Meredith C. McCormack, MD, MHS, Principal Investigator — Johns Hopkins University, Pulmonary and Critical Care Medicine
Locations (1):
- Meredith McCormack, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaviany P, Brigham EP, Collaco JM, Rice JL, Woo H, Wood M, Koehl R, Wu TD, Eakin MN, Koehler K, Hansel NN, McCormack MC. Patterns and predictors of air purifier adherence in children with asthma living in low-income, urban households. J Asthma. 2022 May;59(5):946-955. doi: 10.1080/02770903.2021.1893745. Epub 2021 Mar 10. PMID 33625291